CLINICAL TRIAL: NCT00940498
Title: A Phase 1 Study Of Pf-05212384 (Also Known As Pki-587) Administered As An Intravenous Infusion To Patients With Solid Tumors
Brief Title: Study of PF-05212384 (Also Known as PKI-587)Administered Intravenously To Subjects With Solid Tumors
Acronym: B2151001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: B2151001; 3265K1-1002 (Other: Alias Study Number); 2009-012379-85 (EudraCT Number)
Record Dates: First submitted 2009-07-14; First posted 2009-07-16 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-02

CONDITIONS: Neoplasms
Keywords: Phase 1; Dose Finding; Solid Tumors; Tumors; PF-05212384
MeSH Terms: conditions — Neoplasms | interventions — gedatolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): PF-05212384 (also known as PKI-587)
  Interventions: Drug: PF-05212384 (also known as PKI-587)

INTERVENTIONS:
Drug: PF-05212384 (also known as PKI-587) — Intravenous dosing once weekly infusion

SUMMARY:
This is a two-part study of a compound called PF-05212384 (also known as PKI-587). The purpose of part 1 is to identify the Maximum Tolerated Dose (MTD) of PF-05212384 using a Continual Reassessment Method (CRM). Part 1 will include subjects with any solid tumor. In Part 2 two cohorts will be enrolled. One cohort will assess safety, tolerability and preliminary efficacy in 20 subjects at the MTD and will include subjects with breast cancer, ovarian cancer, endometrial cancer, colorectal cancer renal cancer or glioblastoma (a type of brain tumor). The other cohort will include 5 to 15 subjects with any type of tumor who consent to provide tumor biopsies while participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of any solid tumor
* Incurable cancer, with disease progression following at least 1 therapy with no further standard treatment available in the opinion of the investigator.
* At least 1 evaluable lesion per RECIST criteria

Exclusion Criteria:

* Clinically unstable primary or metastatic CNS tumors
* Subjects with known diabetes
* QTc interval greater than 470 ms.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (6):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Insitute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Tennessee Oncology, PLLC, Nashville, Tennessee
- Hospital General Vall D'Hebron, Barcelona, Spain
- King's College London, London, England, United Kingdom

REFERENCES:
- [Derived] Shapiro GI, Bell-McGuinn KM, Molina JR, Bendell J, Spicer J, Kwak EL, Pandya SS, Millham R, Borzillo G, Pierce KJ, Han L, Houk BE, Gallo JD, Alsina M, Brana I, Tabernero J. First-in-Human Study of PF-05212384 (PKI-587), a Small-Molecule, Intravenous, Dual Inhibitor of PI3K and mTOR in Patients with Advanced Cancer. Clin Cancer Res. 2015 Apr 15;21(8):1888-95. doi: 10.1158/1078-0432.CCR-14-1306. Epub 2015 Feb 4. PMID 25652454
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2151001&StudyName=Study%20of%20PF-05212384%20%28also%20known%20as%20PKI-587%29Administered%20Intravenously%20To%20Subjects%20With%20Solid%20Tumors

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in two parts: Part 1 to determine the maximum tolerated dose (MTD) and Part 2 to confirm the MTD. As per the sponsor's decision, data was reported for the combined population of Part 1 and Part 2 which was considered more informative.
Groups:
- Part 1: PF-05212384 10 mg: PF-05212384 10 mg IV infusion, once weekly in each 28-day cycle until progression of disease, uncontrollable toxicity or a decision by the participant or investigator to discontinue during Part 1 (MTD estimation) of the study.
- Part 1: PF-05212384 21 mg: PF-05212384 21 mg IV infusion, once weekly in each 28-day cycle until progression of disease, uncontrollable toxicity or a decision by the participant or investigator to discontinue during Part 1 (MTD estimation) of the study.
- Part 1: PF-05212384 43 mg: PF-05212384 43 mg IV infusion, once weekly in each 28-day cycle until progression of disease, uncontrollable toxicity or a decision by the participant or investigator to discontinue during Part 1 (MTD estimation) of the study.
- Part 1: PF-05212384 89 mg: PF-05212384 89 mg IV infusion, once weekly in each 28-day cycle until progression of disease, uncontrollable toxicity or a decision by the participant or investigator to discontinue during Part 1 (MTD estimation) of the study.
- Part 1 and 2: PF-05212384 154 mg: PF-05212384 154 mg IV infusion, once weekly in each 28-day cycle until progression of disease, uncontrollable toxicity or a decision by the participant or investigator to discontinue during Part 1 (MTD estimation) and Part 2 (MTD confirmation) of the study.
- Part 1: PF-05212384 222 mg: PF-05212384 222 mg IV infusion, once weekly in each 28-day cycle until progression of disease, uncontrollable toxicity or a decision by the participant or investigator to discontinue during Part 1 (MTD estimation) of the study.
- Part 1: PF-05212384 266 mg: PF-05212384-266 mg IV infusion, once weekly in each 28-day cycle until progression of disease, uncontrollable toxicity or a decision by the participant or investigator to discontinue during Part 1 (MTD estimation) of the study.
- Part 1: PF-05212384 319 mg: PF-05212384-319 mg IV infusion, once weekly in each 28-day cycle until progression of disease, uncontrollable toxicity or a decision by the participant or investigator to discontinue during Part 1 (MTD estimation) of the study.
Period: Overall Study
Arm/Group | Part 1: PF-05212384 10 mg | Part 1: PF-05212384 21 mg | Part 1: PF-05212384 43 mg | Part 1: PF-05212384 89 mg | Part 1 and 2: PF-05212384 154 mg | Part 1: PF-05212384 222 mg | Part 1: PF-05212384 266 mg | Part 1: PF-05212384 319 mg
Started | 4 | 4 | 4 | 4 | 43 | 7 | 8 | 4
Completed | 1 | 3 | 1 | 2 | 34 | 6 | 7 | 3
Not Completed | 3 | 1 | 3 | 2 | 9 | 1 | 1 | 1
Not completed — Death | 2 | 0 | 0 | 1 | 5 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 1
Not completed — Disease Progression | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Not treated due to disease related pain | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Groups:
- Part 1: PF-05212384 10 mg: PF-05212384 10 milligram (mg), intravenous (IV) infusion, once weekly in each 28-day cycle until progression of disease, uncontrollable toxicity or a decision by the participant or investigator to discontinue during Part 1 (MTD estimation) of the study.
- Total: Total of all reporting groups
Arm/Group | Part 1: PF-05212384 10 mg | Part 1: PF-05212384 21 mg | Part 1: PF-05212384 43 mg | Part 1: PF-05212384 89 mg | Part 1 and 2: PF-05212384 154 mg | Part 1: PF-05212384 222 mg | Part 1: PF-05212384 266 mg | Part 1: PF-05212384 319 mg | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 42 | 7 | 8 | 4 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 4 | 4 | 34 | 4 | 7 | 4 | 64
  >=65 years | 0 | 1 | 0 | 0 | 8 | 3 | 1 | 0 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 2 | 20 | 5 | 4 | 4 | 40
  Male | 3 | 1 | 3 | 2 | 22 | 2 | 4 | 0 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to Cycle 14, that were absent before treatment or that worsened relative to pre-treatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline up to Cycle 14 (each cycle is 28 days)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-05212384 10 mg | Part 1: PF-05212384 21 mg | Part 1: PF-05212384 43 mg | Part 1: PF-05212384 89 mg | Part 1 and 2: PF-05212384 154 mg | Part 1: PF-05212384 222 mg | Part 1: PF-05212384 266 mg | Part 1: PF-05212384 319 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 42 | 7 | 8 | 4
Participants
  AEs | 4 | 4 | 4 | 4 | 42 | 7 | 8 | 4
  SAEs | 2 | 1 | 1 | 1 | 16 | 0 | 5 | 2

2. Primary Outcome: Number of Participants With Treatment-Emergent Treatment-Related Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Cycle 14, that were absent before treatment or that worsened relative to pretreatment state. Relatedness to drug was assessed by the investigator. Participants with multiple occurrences of an AE within a category were counted once within the category. AEs included both serious and non-serious adverse events.
Time Frame: Baseline up to Cycle 14 (each cycle is 28 days)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-05212384 10 mg | Part 1: PF-05212384 21 mg | Part 1: PF-05212384 43 mg | Part 1: PF-05212384 89 mg | Part 1 and 2: PF-05212384 154 mg | Part 1: PF-05212384 222 mg | Part 1: PF-05212384 266 mg | Part 1: PF-05212384 319 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 42 | 7 | 8 | 4
Participants
  AEs | 3 | 3 | 4 | 4 | 40 | 7 | 8 | 4
  SAEs | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2

3. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: Criteria for laboratory test abnormality: hematology (hemoglobin [less than {<} 0.8*lower limit of normal {LLN}], platelets [<0.5*LLN or greater than {>} 1.75*upper limit of normal {ULN}], white blood cells [<0.6*LLN or >1.5*ULN], lymphocytes [<0.8*LLN or >1.2*ULN], total neutrophils [<0.8*LLN or >1.2*ULN], basophils, eosinophils, monocytes [>1.2*ULN]); coagulation [partial thromboplastin time, prothrombin (PT), PT international ratio [>1.1*ULN]); liver function (total bilirubin [>1.5*ULN], aspartate aminotransferase, alanine aminotransferase, lactate dehydrogenase, alkaline phosphatase [>0.3*ULN], total protein, albumin [<0.8*LLN or >1.2*ULN]).
Time Frame: Baseline up to Cycle 14 (each cycle is 28 days)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-05212384 10 mg | Part 1: PF-05212384 21 mg | Part 1: PF-05212384 43 mg | Part 1: PF-05212384 89 mg | Part 1 and 2: PF-05212384 154 mg | Part 1: PF-05212384 222 mg | Part 1: PF-05212384 266 mg | Part 1: PF-05212384 319 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 42 | 7 | 8 | 4
Participants | 4 | 3 | 4 | 3 | 41 | 7 | 7 | 4

4. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was defined as any of the following events occurring during the first 28 days of study medication and considered at least possibly-related to study medication: Grade 3 nonhematologic AE (including nausea, vomiting, or diarrhea despite optimal therapy; or greater than or equal to [>=] grade 3 asthenia >2 days; or fasting serum glucose >250 milligrams per deciliter (mg/dL) despite optimal therapy); >=Grade 4 thrombocytopenia; Grade 3 thrombocytopenia with bleeding; Grade 4 neutropenia lasting more than 7 days; Febrile neutropenia; other Grade 4 hematologic AE; delay of treatment >2 consecutive weeks due to toxicity. Grades were based on National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: Baseline up to Day 28
Population: DLT evaluable analysis set included all enrolled participants who started treatment and did not have had a major treatment deviation in the first cycle of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-05212384 10 mg | Part 1: PF-05212384 21 mg | Part 1: PF-05212384 43 mg | Part 1: PF-05212384 89 mg | Part 1 and 2: PF-05212384 154 mg | Part 1: PF-05212384 222 mg | Part 1: PF-05212384 266 mg | Part 1: PF-05212384 319 mg
Number analyzed (Participants) | 3 | 4 | 3 | 4 | 40 | 7 | 8 | 4
Participants | 0 | 0 | 0 | 0 | 2 | 5 | 3 | 2

5. Primary Outcome: Recommended Phase-2 Dose (RP2D)
Description: RP2D of PF-05212384 was determined based on the safety profile including laboratory and clinical assessments and pharmacodynamics findings.
Time Frame: Baseline up to Cycle 14 (each cycle is 28 days)
Population: Safety analysis population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: mg
Groups:
- PF-05212384 : All Participants: All participants who received PF-05212384 10 mg or 21 mg or 43 mg or 89 mg or 154 mg or 222 mg or 266 mg or 319 mg, intravenous infusion, once weekly in each 28 day cycle until progression of disease, uncontrollable toxicity, or a decision by the participant or investigator to discontinue.
Arm/Group | PF-05212384 : All Participants
Number analyzed (Participants) | 77
mg | 154

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-05212384: Single and Multiple Dose
Time Frame: Cycle 1: predose, 0.5, 2, 3, 6, 24, 72, 120 and 168 hours postdose on Day 1; Cycle 2: predose, 0.5, 24, 72, 120 hours postdose on Day 1
Population: PK parameter analysis population included all enrolled participants who received at least 1 dose of study drug and had at least 1 of the PK parameters of interest estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1: PF-05212384 10 mg | Part 1: PF-05212384 21 mg | Part 1: PF-05212384 43 mg | Part 1: PF-05212384 89 mg | Part 1 and 2: PF-05212384 154 mg | Part 1: PF-05212384 222 mg | Part 1: PF-05212384 266 mg | Part 1: PF-05212384 319 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 42 | 7 | 8 | 3
nanogram per milliliter (ng/mL)
  Cycle 1 | 714.1 (33) | 1674 (10) | 3317 (10) | 6508 (106) | 9988 (28) | 14730 (54) | 14240 (29) | 27090 (26)
  Cycle 2: number analyzed (Participants) | 3 | 3 | 4 | 4 | 31 | 4 | 7 | 2
  Cycle 2 | 542.8 (28) | 1482 (24) | 2601 (33) | 4250 (43) | 8594 (64) | 15660 (86) | 10840 (46) | NA (NA) — Results were not summarized if evaluable participants were less than 3, considered as insufficient values by investigator to calculate a reliable estimation.

7. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-05212384: Single Dose
Description: Area under the plasma concentration versus time curve from time zero (predose) to time of last quantifiable concentration (Clast).
Time Frame: Cycle 1: predose, 0.5, 2, 3, 6, 24, 72, 120 and 168 hours postdose on Day 1
Population: PK parameter analysis population included all enrolled participants who received at least 1 dose of study drug and had at least 1 of the PK parameters of interest estimated. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter(ng*hr/mL)
Arm/Group | Part 1: PF-05212384 10 mg | Part 1: PF-05212384 21 mg | Part 1: PF-05212384 43 mg | Part 1: PF-05212384 89 mg | Part 1 and 2: PF-05212384 154 mg | Part 1: PF-05212384 222 mg | Part 1: PF-05212384 266 mg | Part 1: PF-05212384 319 mg
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 42 | 7 | 8 | 3
nanogram*hour per milliliter(ng*hr/mL) | 1149 (35) | 2367 (24) | 5741 (14) | 13090 (77) | 15780 (28) | 26550 (30) | 28180 (36) | 46760 (2)

8. Secondary Outcome: Plasma Decay Half-Life (t1/2) of PF-05212384: Single and Multiple Dose
Description: Plasma decay half-life is the time measured for the plasma concentration of drug to decrease by one half.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours (hr)
Arm/Group | Part 1: PF-05212384 10 mg | Part 1: PF-05212384 21 mg | Part 1: PF-05212384 43 mg | Part 1: PF-05212384 89 mg | Part 1 and 2: PF-05212384 154 mg | Part 1: PF-05212384 222 mg | Part 1: PF-05212384 266 mg | Part 1: PF-05212384 319 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 42 | 7 | 8 | 3
hours (hr)
  Cycle 1: number analyzed (Participants) | 4 | 4 | 3 | 4 | 39 | 6 | 7 | 3
  Cycle 1 | 15.14 (6.1475) | 17.34 (9.8683) | 40.73 (7.7822) | 35.95 (9.1267) | 35.84 (6.2454) | 33.33 (4.8144) | 37.51 (4.8516) | 38.53 (4.5457)
  Cycle 2: number analyzed (Participants) | 0 | 1 | 2 | 3 | 23 | 4 | 6 | 1
  Cycle 2 |  | NA (NA) — Results were not summarized if evaluable participants were less than 3, considered as insufficient values by investigator to calculate a reliable estimation. | NA (NA) — Results were not summarized if evaluable participants were less than 3, considered as insufficient values by investigator to calculate a reliable estimation. | 37.10 (4.4238) | 35.97 (5.3197) | 34.03 (6.6385) | 36.38 (5.1188) | NA (NA) — Results were not summarized if evaluable participants were less than 3, considered as insufficient values by investigator to calculate a reliable estimation.

9. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of PF-05212384: Single Dose
Description: AUCinf= Area under the plasma concentration versus time curve (AUC) from time zero (predose) to extrapolated infinite time (0 - inf).
Time Frame: Cycle 1: predose, 0.5, 2, 3, 6, 24, 72, 120 and 168 hours postdose on Day 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1: PF-05212384 10 mg | Part 1: PF-05212384 21 mg | Part 1: PF-05212384 43 mg | Part 1: PF-05212384 89 mg | Part 1 and 2: PF-05212384 154 mg | Part 1: PF-05212384 222 mg | Part 1: PF-05212384 266 mg | Part 1: PF-05212384 319 mg
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 39 | 6 | 7 | 3
ng*hr/mL | 1238 (32) | 2485 (23) | 5881 (14) | 13280 (78) | 16250 (28) | 27210 (33) | 28280 (39) | 47460 (2)

10. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-05212384: Single and Multiple Dose
Description: Area under the concentration curve from time 0 to end of dosing interval (AUCtau), where dosing interval was 168 hours (1 Week). For Cycle 2, the last PK sample for parameter calculations was on 120 hours after the Day 1 dose, however AUCtau was extrapolated to 168 hours using t1/2.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1: PF-05212384 10 mg | Part 1: PF-05212384 21 mg | Part 1: PF-05212384 43 mg | Part 1: PF-05212384 89 mg | Part 1 and 2: PF-05212384 154 mg | Part 1: PF-05212384 222 mg | Part 1: PF-05212384 266 mg | Part 1: PF-05212384 319 mg
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 42 | 7 | 8 | 3
ng*hr/mL
  Cycle 1 | 1256 (29) | 2604 (22) | 5753 (13) | 13100 (78) | 15810 (28) | 26740 (30) | 28220 (36) | 46730 (2)
  Cycle 2: number analyzed (Participants) | 3 | 2 | 3 | 3 | 23 | 4 | 6 | 1
  Cycle 2 | 2991 (26) | NA (NA) — Results were not summarized if evaluable participants were less than 3, considered as insufficient values by investigator to calculate a reliable estimation. | 15820 (29) | 25010 (49) | 47130 (54) | 79380 (64) | 61910 (42) | NA (NA) — Results were not summarized if evaluable participants were less than 3, considered as insufficient values by investigator to calculate a reliable estimation.

11. Secondary Outcome: Number of Participants With Maximum Increase From Baseline in Corrected QT Interval
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. The time corresponding to beginning of depolarization to repolarization of the ventricles (QT interval) was adjusted for RR interval using QT and RR from each ECG by Fridericia's formula (QTcF = QT divided by cube root of RR) and by Bazette's formula (QTcB = QT divided by square root of RR). Number of Participants with maximum increase from baseline in QTcB and QTcF of < 30 msec, between <=30 to <60 msec and >=60 were reported.
Time Frame: Baseline up to Cycle 14 (each cycle is 28 days)
Population: The QTc analysis set included all enrolled participants who had at least one ECG assessment after receiving PF-05212384
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-05212384 10 mg | Part 1: PF-05212384 21 mg | Part 1: PF-05212384 43 mg | Part 1: PF-05212384 89 mg | Part 1 and 2: PF-05212384 154 mg | Part 1: PF-05212384 222 mg | Part 1: PF-05212384 266 mg | Part 1: PF-05212384 319 mg
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 42 | 7 | 8 | 4
Participants
  QTcB: Change <30 | 3 | 3 | 3 | 3 | 26 | 6 | 4 | 4
  QTcB: <= 30 and <60 | 1 | 1 | 1 | 0 | 13 | 1 | 3 | 0
  QTcB: Change >=60 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0
  QTcF: Change <30 | 3 | 3 | 4 | 3 | 34 | 6 | 6 | 4
  QTcF: <= 30 and <60 | 1 | 1 | 0 | 0 | 7 | 1 | 2 | 0
  QTcF: Change >=60 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

12. Secondary Outcome: Change From Baseline in Serum Glucose at Day 2 of Cycle 1, Day 1 of Cycle 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and End of Treatment
Time Frame: Baseline, Day 2 of Cycle 1, thereafter Day 1 of Cycle 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 (each cycle 28 days) , end of treatment visit (up to Cycle 14)
Population: Serum biomarker analysis set included all enrolled participants who started treatment and had baseline and on-treatment serum biomarker samples successfully analyzed for at least 1 biomarker.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Part 1: PF-05212384 10 mg | Part 1: PF-05212384 21 mg | Part 1: PF-05212384 43 mg | Part 1: PF-05212384 89 mg | Part 1 and 2: PF-05212384 154 mg | Part 1: PF-05212384 222 mg | Part 1: PF-05212384 266 mg | Part 1: PF-05212384 319 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 41 | 7 | 7 | 4
milligram per deciliter (mg/dL)
  Baseline: number analyzed (Participants) | 4 | 4 | 4 | 4 | 38 | 5 | 4 | 3
  Baseline | 100.3 (14.15) | 103.1 (14.55) | 87.0 (6.22) | 91.1 (7.40) | 95.6 (13.48) | 96.7 (10.85) | 88.4 (18.14) | 93.3 (3.06)
  Change at Cycle 1 Day 2: number analyzed (Participants) | 4 | 2 | 3 | 3 | 40 | 7 | 7 | 4
  Change at Cycle 1 Day 2 | 12.5 (29.59) | -4.0 (7.07) | 0.3 (10.60) | 13.5 (4.08) | 13.7 (21.49) | 21.1 (24.97) | 65.5 (41.41) | 54.5 (94.71)
  Change at Cycle 2 Day 1: number analyzed (Participants) | 3 | 4 | 4 | 4 | 33 | 5 | 6 | 2
  Change at Cycle 2 Day 1 | 1.0 (18.36) | 28.4 (26.90) | 11.5 (7.59) | 3.0 (9.56) | 2.8 (15.74) | 5.0 (6.67) | 12.9 (14.45) | 9.5 (3.54)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 2 | 14 | 2 | 5 | 2
  Change at Cycle 3 Day 1 | 19.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 19.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 2.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 9.3 (4.68) | 10.4 (29.02) | 16.0 (15.56) | 26.9 (33.77) | -11.0 (1.41)
  Change at Cycle 4 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 2 | 8 | 1 | 4 | 2
  Change at Cycle 4 Day 1 | -1.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 7.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 3.6 (7.64) | 2.0 (10.81) | 26.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 41.6 (45.85) | 6.5 (0.71)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 1 | 1 | 0 | 2 | 5 | 1 | 4 | 2
  Change at Cycle 5 Day 1 | -9.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 8.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  | 8.2 (8.78) | -3.8 (9.39) | -3.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 29.7 (33.08) | -7.0 (2.83)
  Change at Cycle 6 Day 1: number analyzed (Participants) | 1 | 1 | 0 | 2 | 3 | 1 | 4 | 2
  Change at Cycle 6 Day 1 | -7.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 2.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  | 1.0 (1.41) | -10.0 (8.66) | 14.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 29.1 (28.17) | 5.0 (5.66)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2 | 0 | 4 | 1
  Change at Cycle 7 Day 1 | -9.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 10.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  | 8.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -5.0 (2.83) |  | 48.7 (50.13) | 7.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at Cycle 8 Day 1: number analyzed (Participants) | 1 | 1 | 0 | 1 | 2 | 0 | 3 | 1
  Change at Cycle 8 Day 1 | -12.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 6.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  | 11.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 1.5 (21.92) |  | 39.0 (32.70) | -3.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at Cycle 9 Day 1: number analyzed (Participants) | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 1
  Change at Cycle 9 Day 1 | -7.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 9.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  | 5.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  |  | 65.0 (42.66) | 1.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at Cycle 10 Day 1: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Change at Cycle 10 Day 1 | -2.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 15.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  |  |  |  |  | 11.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at Cycle 11 Day 1: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Change at Cycle 11 Day 1 | -8.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -15.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  |  |  |  | 39.6 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  Change at Cycle 12 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Change at Cycle 12 Day 1 | -9.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  |  |  |  |  | 28.8 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  Change at Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Change at Cycle 13 Day 1 |  |  |  |  |  |  | -1.8 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  Change at Cycle 14 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Change at Cycle 14 Day 1 |  |  |  |  |  |  | 36.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  Change at EOT: number analyzed (Participants) | 3 | 3 | 4 | 3 | 29 | 6 | 7 | 2
  Change at EOT | 10.7 (34.12) | 7.2 (12.64) | 23.3 (31.48) | 16.1 (15.07) | 7.4 (21.08) | -6.7 (13.52) | 27.5 (32.75) | 42.0 (72.12)

13. Secondary Outcome: Change From Baseline in Serum Insulin at Day 2 of Cycle 1, Day 1 of Cycle 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and End of Treatment
Time Frame: as for outcome 12
Population: Serum biomarker analysis set. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure (OM).
Measure: Mean (Standard Deviation); unit: microunits per milliliter (mcU/mL)
Arm/Group | Part 1: PF-05212384 10 mg | Part 1: PF-05212384 21 mg | Part 1: PF-05212384 43 mg | Part 1: PF-05212384 89 mg | Part 1 and 2: PF-05212384 154 mg | Part 1: PF-05212384 222 mg | Part 1: PF-05212384 266 mg | Part 1: PF-05212384 319 mg
Number analyzed (Participants) | 4 | 1 | 3 | 2 | 37 | 6 | 7 | 4
microunits per milliliter (mcU/mL)
  Baseline ( n=4,1,3,2,35,4,4,3): number analyzed (Participants) | 4 | 1 | 3 | 2 | 35 | 4 | 4 | 3
  Baseline ( n=4,1,3,2,35,4,4,3) | 23.8 (22.90) | 10.2 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 8.6 (4.40) | 5.3 (1.84) | 13.1 (9.34) | 18.2 (14.14) | 5.9 (7.86) | 11.4 (7.00)
  Change at Cycle 1 Day 2 (n =4,1,3,2,37,6,7,4) | 4.0 (33.56) | 2.5 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 2.9 (6.81) | 4.7 (2.90) | 22.8 (25.68) | 40.9 (47.05) | 57.5 (41.66) | 110.3 (117.23)
  Change at Cycle 2 Day 1 (n =0,0,0,2,27,5,3,1): number analyzed (Participants) | 0 | 0 | 0 | 2 | 27 | 5 | 3 | 1
  Change at Cycle 2 Day 1 (n =0,0,0,2,27,5,3,1) |  |  |  | 5.4 (3.54) | 1.3 (8.66) | 2.6 (7.88) | 7.3 (10.31) | -2.9 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at Cycle 3 Day 1 (n =0,1,1,1,14,1,3,1): number analyzed (Participants) | 0 | 1 | 1 | 1 | 14 | 1 | 3 | 1
  Change at Cycle 3 Day 1 (n =0,1,1,1,14,1,3,1) |  | 1.4 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 2.1 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.9 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -0.7 (11.66) | 4.2 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 2.1 (4.38) | 18.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at Cycle 4 Day 1 (n =0,0,1,1,8,0,3,2): number analyzed (Participants) | 0 | 0 | 1 | 1 | 8 | 0 | 3 | 2
  Change at Cycle 4 Day 1 (n =0,0,1,1,8,0,3,2) |  |  | 3.1 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 3.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 2.9 (6.35) |  | 4.2 (2.54) | 0.6 (3.32)
  Change at Cycle 5 Day 1 (n =0,1,0,1,5,0,3,1): number analyzed (Participants) | 0 | 1 | 0 | 1 | 5 | 0 | 3 | 1
  Change at Cycle 5 Day 1 (n =0,1,0,1,5,0,3,1) |  | -0.7 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  | 0.1 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 2.3 (5.24) |  | 3.3 (1.86) | -3.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C6D1 (n=0,1,0,1,3,0,2,2): number analyzed (Participants) | 0 | 1 | 0 | 1 | 3 | 0 | 2 | 2
  Change at C6D1 (n=0,1,0,1,3,0,2,2) |  | -1.2 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  | 3.1 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.9 (5.14) |  | 0.8 (0.07) | 0.3 (0.42)
  Change at Cycle 7 Day 1 (n=0,1,0,1,2,0,3,1): number analyzed (Participants) | 0 | 1 | 0 | 1 | 2 | 0 | 3 | 1
  Change at Cycle 7 Day 1 (n=0,1,0,1,2,0,3,1) |  | 0.9 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  | 0.2 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 2.1 (0.85) |  | 6.9 (8.31) | 5.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at Cycle 8 Day 1 (n =0,1,0,1,2,0,3,1): number analyzed (Participants) | 0 | 1 | 0 | 1 | 2 | 0 | 3 | 1
  Change at Cycle 8 Day 1 (n =0,1,0,1,2,0,3,1) |  | -1.9 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  | 3.1 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 4.5 (4.17) |  | -0.9 (2.71) | -1.4 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at Cycle 9 Day 1 ( n=0,1,0,1,0,0,2,1): number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1
  Change at Cycle 9 Day 1 ( n=0,1,0,1,0,0,2,1) |  | 5.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  | 0.9 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  |  | 1.8 (4.60) | -1.7 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at Cycle 10 Day 1 (n =1,1,0,0,0,0,0,1): number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Change at Cycle 10 Day 1 (n =1,1,0,0,0,0,0,1) | -18.3 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 3.4 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  |  |  |  |  | 5.8 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at Cycle 11 Day 1 (n =1,1,0,0,0,0,1,0): number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Change at Cycle 11 Day 1 (n =1,1,0,0,0,0,1,0) | -32.2 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.1 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  |  |  |  | 38.6 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  Change at Cycle 12 Day 1 (n =1,0,0,0,0,0,0,0): number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Change at Cycle 12 Day 1 (n =1,0,0,0,0,0,0,0) | -4.3 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  |  |  |  |  |  |
  Change at Cycle 13 D 1 (n =0,0,0,0,0,0,1,0): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Change at Cycle 13 D 1 (n =0,0,0,0,0,0,1,0) |  |  |  |  |  |  | 22.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  Change at Cycle 14 Day 1 (n =0,0,0,0,0,0,1,0): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Change at Cycle 14 Day 1 (n =0,0,0,0,0,0,1,0) |  |  |  |  |  |  | 107.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  Change at EOT (n =1,0,1,1,21,4,6,1): number analyzed (Participants) | 1 | 0 | 1 | 1 | 21 | 4 | 6 | 1
  Change at EOT (n =1,0,1,1,21,4,6,1) | 19.1 (NA) — Standard deviation was not estimable since only one participant was evaluable. |  | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.8 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 1.7 (8.59) | -4.8 (9.04) | 19.6 (21.67) | -4.3 (NA) — Standard deviation was not estimable since only one participant was evaluable.

14. Secondary Outcome: Change From Baseline in Serum C-peptide at Day 2 of Cycle 1, Day 1 of Cycle 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and End of Treatment
Time Frame: as for outcome 12
Population: Serum biomarker analysis set. Here, N= participants evaluable for this outcome measure. Data for this outcome measure was not planned to be analyzed for reporting arms: PF-05212384 10 mg, 21 mg, 43 mg, 89 mg, and 319 mg, as pre specified in protocol Amendment 5.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1 and 2: PF-05212384 154 mg | Part 1: PF-05212384 222 mg | Part 1: PF-05212384 266 mg
Number analyzed (Participants) | 35 | 5 | 3
ng/mL
  Baseline | 3.0 (1.82) | 3.0 (1.19) | 4.6 (1.92)
  Change at Cycle 1 Day 2: number analyzed (Participants) | 34 | 5 | 2
  Change at Cycle 1 Day 2 | 3.6 (2.23) | 6.2 (4.23) | 5.0 (5.37)
  Change at Cycle 2 Day 1: number analyzed (Participants) | 26 | 4 | 2
  Change at Cycle 2 Day 1 | 0.4 (1.36) | 1.0 (1.30) | -1.1 (2.23)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 12 | 1 | 2
  Change at Cycle 3 Day 1 | 0.5 (1.15) | 2.5 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -1.8 (3.11)
  Change at Cycle 4 Day 1: number analyzed (Participants) | 7 | 0 | 2
  Change at Cycle 4 Day 1 | 0.9 (1.45) |  | 0.1 (1.56)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 4 | 0 | 2
  Change at Cycle 5 Day 1 | 0.4 (0.86) |  | -1.2 (2.87)
  Change at Cycle 6 Day 1: number analyzed (Participants) | 2 | 0 | 2
  Change at Cycle 6 Day 1 | -0.0 (0.54) |  | -0.3 (1.60)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 2 | 0 | 2
  Change at Cycle 7 Day 1 | 0.1 (0.36) |  | 1.9 (1.20)
  Change at Cycle 8 Day 1: number analyzed (Participants) | 2 | 0 | 2
  Change at Cycle 8 Day 1 | 0.3 (0.14) |  | -0.9 (3.75)
  Change at Cycle 9 Day 1: number analyzed (Participants) | 0 | 0 | 1
  Change at Cycle 9 Day 1 |  |  | 2.9 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 0
  Change at Cycle 11 Day 1: number analyzed (Participants) | 0 | 0 | 0
  Change at Cycle 12 Day 1: number analyzed (Participants) | 0 | 0 | 0
  Change at Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 0
  Change at Cycle 14 Day 1: number analyzed (Participants) | 0 | 0 | 0
  Change at EOT: number analyzed (Participants) | 24 | 5 | 2
  Change at EOT | 1.1 (1.82) | -0.1 (0.80) | 5.3 (1.68)

15. Secondary Outcome: Change From Baseline in Hair Follicle Biopsy Biomarkers at Cycle 1 Day 1
Description: Analysis of hair follicles was conducted using a Reverse Phase Microarrays (RPMA) assay. Phosphoprotein biomarkers measured were pAkt S473, pAkt T308, pStat3 (Y705), Ki-67, and pPRAS40 (T246).
Time Frame: Baseline, 2, 3 and 72 hours (H) postdose on Day 1 of Cycle 1
Population: Hair follicle analysis set. Here, N= participants evaluable for this outcome measure. Data for this outcome measure was not planned to be analyzed for reporting arms: PF-05212384 10 mg, 21 mg, 43 mg, 89 mg, and 319 mg, as pre specified in protocol Amendment 5.
Measure: Mean (Standard Deviation); unit: normalized fluorescence units (NFU)
Arm/Group | Part 1 and 2: PF-05212384 154 mg | Part 1: PF-05212384 222 mg | Part 1: PF-05212384 266 mg
Number analyzed (Participants) | 20 | 4 | 1
normalized fluorescence units (NFU)
  Baseline: pAkt S473: number analyzed (Participants) | 19 | 4 | 0
  Baseline: pAkt S473 | 12.2 (4.58) | 17.2 (5.26) |
  Baseline: pAkt T308: number analyzed (Participants) | 20 | 3 | 0
  Baseline: pAkt T308 | 44.3 (19.41) | 36.2 (15.95) |
  Baseline: pStat3 (Y705): number analyzed (Participants) | 17 | 2 | 0
  Baseline: pStat3 (Y705) | 172.3 (47.26) | 224.2 (117.43) |
  Baseline: Ki-67: number analyzed (Participants) | 19 | 3 | 1
  Baseline: Ki-67 | 82.1 (21.79) | 128.1 (30.80) | 145.7 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Baseline: pPRAS40 (T246): number analyzed (Participants) | 19 | 3 | 0
  Baseline: pPRAS40 (T246) | 111.7 (31.75) | 99.6 (30.11) |
  Change at C1D1 2H:pAkt S473: number analyzed (Participants) | 18 | 3 | 0
  Change at C1D1 2H:pAkt S473 | -1.7 (3.59) | 6.8 (5.77) |
  Change at C1D1 2H:pAkt T308: number analyzed (Participants) | 18 | 1 | 0
  Change at C1D1 2H:pAkt T308 | 2.3 (17.06) | -4.6 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  Change at C1D1 2H:pStat3 (Y705): number analyzed (Participants) | 15 | 1 | 0
  Change at C1D1 2H:pStat3 (Y705) | -6.2 (34.78) | 126.3 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  Change at C1D1 2H:Ki-67: number analyzed (Participants) | 15 | 1 | 1
  Change at C1D1 2H:Ki-67 | 1.0 (29.41) | 34.7 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -36.2 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Change at C1D1 2H:pPRAS40-T246: number analyzed (Participants) | 15 | 3 | 0
  Change at C1D1 2H:pPRAS40-T246 | -27.4 (22.59) | 42.0 (26.01) |
  Change at C1D1 3hr: pAkt S473: number analyzed (Participants) | 15 | 4 | 0
  Change at C1D1 3hr: pAkt S473 | -0.9 (2.93) | 0.2 (9.26) |
  Change at C1D1 3hr: pAkt T308: number analyzed (Participants) | 16 | 3 | 0
  Change at C1D1 3hr: pAkt T308 | 0.4 (14.25) | 6.9 (18.50) |
  Change at C1D1 3H: pStat3 (Y705): number analyzed (Participants) | 11 | 1 | 0
  Change at C1D1 3H: pStat3 (Y705) | -11.7 (54.88) | -142.2 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  Change at C1D1 3hr: Ki-67: number analyzed (Participants) | 13 | 2 | 0
  Change at C1D1 3hr: Ki-67 | -8.5 (23.59) | 25.2 (15.68) |
  Change at C1D1 3H:pPRAS40-T246: number analyzed (Participants) | 12 | 3 | 0
  Change at C1D1 3H:pPRAS40-T246 | -27.8 (27.11) | 49.8 (56.37) |
  Change at C1D4 72H:pAkt S473: number analyzed (Participants) | 12 | 3 | 0
  Change at C1D4 72H:pAkt S473 | -0.9 (3.69) | 1.7 (9.45) |
  Change at C1D4 72H:pAkt-T308: number analyzed (Participants) | 13 | 3 | 0
  Change at C1D4 72H:pAkt-T308 | 9.4 (38.19) | 11.8 (15.16) |
  Change at C1D4 72H: pStat3 (Y705): number analyzed (Participants) | 9 | 1 | 0
  Change at C1D4 72H: pStat3 (Y705) | 1.9 (35.99) | 239.8 (NA) — Standard deviation was not estimable since only one participant was evaluable. |
  Change at C1D4 72hr: Ki-67: number analyzed (Participants) | 9 | 3 | 0
  Change at C1D4 72hr: Ki-67 | 5.7 (38.59) | 13.5 (57.80) |
  Change atC1D4-72H:pPRAS40 T246: number analyzed (Participants) | 13 | 2 | 0
  Change atC1D4-72H:pPRAS40 T246 | -2.1 (31.55) | 35.6 (77.10) |

16. Secondary Outcome: Change From Baseline in Fresh Tumor Biopsy Biomarkers at Cycle 1 Day 22
Description: Tumor biopsies were taken from participants of reporting arm PF-05212384 154 mg dose level at baseline and at Cycle 1/Day 22. Biopsies were fixed in optimal cutting temperature compound and analyzed via RPMA. The biomarkers tested were phosphorylated versions of the proteins: AKT S473, AKT T308, FKHR T24 / FKHR1 T32, and STAT3. This outcome measure was planned to be analyzed only for the reporting arm Part 1 and 2: PF-05212384 154 mg, as pre-specified in protocol.
Time Frame: Baseline, Day 22 of Cycle 1
Population: Tumor biopsy analysis set=all enrolled participants who had treatment &had baseline,on-treatment tumor tissue successfully analyzed for at least 1 biomarker.N=participants evaluable for this OM. This OM was planned to analyzed only in reporting arm- Part 1 and 2:PF-05212384 154 mg.
Measure: Mean (Standard Deviation); unit: normalized to cytokeratin (NFC)
Arm/Group | Part 1 and 2: PF-05212384 154 mg
Number analyzed (Participants) | 8
normalized to cytokeratin (NFC)
  Baseline: AKT S473 | 34.3 (26.82)
  Baseline: AKT T308: number analyzed (Participants) | 7
  Baseline: AKT T308 | 38.5 (25.80)
  Baseline: FKHR T24 / FKHR1 T32 | 145.1 (113.99)
  Baseline: STAT3: number analyzed (Participants) | 7
  Baseline: STAT3 | 231.4 (219.22)
  Change at C1D22: AKT S473 | -12.3 (36.88)
  Change at C1D22: AKT T308: number analyzed (Participants) | 7
  Change at C1D22: AKT T308 | -5.8 (25.42)
  Change at C1D22: FKHR T24 / FKHR1 T32 | -27.0 (82.92)
  Change at C1D22: STAT3: number analyzed (Participants) | 7
  Change at C1D22: STAT3 | -45.6 (139.67)

17. Secondary Outcome: Number of Participants With Mutation, Deletion, Amplification in Phosphatidylinositol 3-kinase (PI3K) Pathway Signaling Related Genes and/or Proteins in Biopsied Tumor Tissue
Description: Biopsied tumor tissue was analyzed for alterations in the phosphoinositide-3-kinase/rat sarcoma (PI3K/RAS) signaling pathway by molecular approaches. The biomarkers studied were PIK3CA and phosphatase and tensin homolog (PTEN) by immunohistochemistry.
Time Frame: Baseline
Population: Baseline tumor tissue biomarker analysis set: All enrolled patients who start treatment and had baseline tumor tissues successfully analyzed for at least one of the biomarkers. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- PF-05212384 : All Participants: PF-05212384-10,21,43,89,154,222,266,319 milligram (mg) intravenous infusion over approximately 30 minutes once weekly in each 28 day cycle until progression of disease, uncontrollable toxicity, or a decision by the patient or investigator to discontinue.
Arm/Group | PF-05212384 : All Participants
Number analyzed (Participants) | 70
Participants
  PTEN Mutation: Present | NA — Data for mutation was not collected based on sponsors decision since it was not a biologically relevant parameter for PTEN.
  PTEN Mutation: Absent | NA — Data for mutation was not collected based on sponsors decision since it was not a biologically relevant parameter for PTEN.
  PTEN Deletion: Present | 28
  PTEN Deletion: Absent | 28
  PTEN Amplification: Present | NA — Data for amplification was not collected based on sponsors decision since it was not a biologically relevant parameter for PTEN.
  PTEN Amplification: Absent | NA — Data for amplification was not collected based on sponsors decision since it was not a biologically relevant parameter for PTEN.
  PIK3CA Mutation: Present | 4
  PIK3CA Mutation: Absent | 27
  PIK3CA Deletion: Present | NA — Data for deletion was not collected based on sponsors decision since it was not a biologically relevant parameter for PIK3CA.
  PIK3CA Deletion: Absent | NA — Data for deletion was not collected based on sponsors decision since it was not a biologically relevant parameter for PIK3CA.
  PIK3CA Amplification: Present | 2
  PIK3CA Amplification: Absent | 56

18. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Objective response was defined as having complete response (CR) or Partial Response (PR) assessed by RECIST 1.1. CR was defined as disappearance of all target, non-target lesions; normalization of tumor marker level and all lymph nodes size was <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters). Percentage of participants with objective response were reported.
Time Frame: Baseline until disease progression or death due to any cause (up to Cycle 14 [each cycle 28 days])
Population: Response-evaluable population included participants who received at least 1 dose of study drug, had an adequate baseline tumor assessment and at least 1 post baseline disease assessment for analyses of response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- PF-05212384 : All Participants: Entire study population treated with PF-05212384-10,21,43,89,154,222,266,319 mg intravenous infusion over approximately 30 minutes once weekly in each 28 day cycle until progression of disease, uncontrollable toxicity, or a decision by the participant or investigator to discontinue.
Arm/Group | PF-05212384 : All Participants
Number analyzed (Participants) | 77
percentage of participants | 2.6 [0.3 to 9.1]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Part 1: PF-05212384 10 mg | Part 1: PF-05212384 21 mg | Part 1: PF-05212384 43 mg | Part 1: PF-05212384 89 mg | Part 1 and 2: PF-05212384 154 mg | Part 1: PF-05212384 222 mg | Part 1: PF-05212384 266 mg | Part 1: PF-05212384 319 mg
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/4 | 1/4 | 1/4 | 16/42 | 0/7 | 5/8 | 2/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 4/4 | 4/4 | 42/42 | 7/7 | 8/8 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: PF-05212384 10 mg (N=4) | Part 1: PF-05212384 21 mg (N=4) | Part 1: PF-05212384 43 mg (N=4) | Part 1: PF-05212384 89 mg (N=4) | Part 1 and 2: PF-05212384 154 mg (N=42) | Part 1: PF-05212384 222 mg (N=7) | Part 1: PF-05212384 266 mg (N=8) | Part 1: PF-05212384 319 mg (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 2 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aortic disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: PF-05212384 10 mg (N=4) | Part 1: PF-05212384 21 mg (N=4) | Part 1: PF-05212384 43 mg (N=4) | Part 1: PF-05212384 89 mg (N=4) | Part 1 and 2: PF-05212384 154 mg (N=42) | Part 1: PF-05212384 222 mg (N=7) | Part 1: PF-05212384 266 mg (N=8) | Part 1: PF-05212384 319 mg (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 6 | 1 | 2 | 2
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 6 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 3 | 3 | 2 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 13 | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 9 | 2 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastric varices (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gingival inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 2 | 2 | 1 | 22 | 3 | 6 | 3
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Painful defaecation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2
Perianal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Rectal discharge (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 5 | 2 | 2 | 1
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 15 | 2 | 5 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 14 | 1 | 4 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 1
Early satiety (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 2 | 2 | 0 | 10 | 3 | 3 | 2
Feeling jittery (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 1 | 0 | 19 | 5 | 6 | 3
Oedema peripheral (General disorders) | 2 | 1 | 0 | 0 | 2 | 0 | 1 | 1
Pain (General disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 1 | 11 | 1 | 2 | 1
Sensation of foreign body (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Lip infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 0 | 2 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sputum purulent (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 0 | 9 | 2 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 10 | 2 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 0 | 1 | 0 | 6 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Liver palpable subcostal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatic enzymes increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 2 | 1 | 16 | 3 | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 4 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 12 | 1 | 4 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 3 | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 3 | 2 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 4 | 0 | 1 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 9 | 0 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 3 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 4 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 8 | 2 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 4 | 1 | 1 | 0
Hemianopia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Motor dysfunction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 6 | 1 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Renal vein thrombosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scrotal swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 9 | 2 | 4 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 5 | 3 | 3 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 4 | 1 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peau d'orange (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 4 | 0 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | 6 | 0 | 6 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.